CLINICAL TRIAL: NCT04784494
Title: Magnetic Seizure Therapy for Parkinson's Disease
Brief Title: MST for Parkinson's Disease
Acronym: MST-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-01049
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease; Depression; Movement Disorders; Major Depressive Disorder
Keywords: Magnetic Seizure Therapy; MST; Convulsive Therapy
MeSH Terms: conditions — Parkinson Disease; Depression; Movement Disorders; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magnetic Seizure Therapy (Experimental): MST treatments will be administered using the MagPro XP MST with Cool TwinCoil.
  Interventions: Device: Magnetic Seizure Theapy (MagPro XP MST)

INTERVENTIONS:
Device: Magnetic Seizure Theapy (MagPro XP MST) — MST treatment will be administered over the frontal/vertex cortex using 100 Hz stimulation using the MagPro XP MST with Cool TwinCoil. The MST determination of seizure threshold will be done using 100% machine output applied at 100 Hz at progressively escalating train durations, commencing at 2 seconds and increasing by 2 seconds with each subsequent stimulation until an adequate seizure is produced. During subsequent sessions, one stimulation will be delivered using a train duration that is 4 seconds longer than the train duration at threshold (with a maximum train duration of 10 seconds).
  MST treatments will be administered twice a week, for up to 16 treatments. This will be performed under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes.
  Other Names: MagPro MST (Tonica Elektronik A/S, Denmark)

SUMMARY:
This trial aims to test the feasibility of Magnetic Seizure Therapy (MST) for Depression in patients diagnosed with Parkinson's Disease.

DETAILED DESCRIPTION:
This is a phase II, single-arm open-label feasibility trial testing the feasibility of MST for dPD. The trial will occur over 18 months at one academic center in Canada (UBC). The enrollment goal is 20 patients with Parkinson's disease and comorbid moderate/severe depression. Research subjects will provide informed consent before enrollment and participation in any research procedures.The study design follows international CONSORT guidelines for the reporting of results in feasibility trials.

Treatment will be administered two days per week (Tuesday/Thursday). This frequency has been chosen as research indicates that depression outcomes at the end of a course of ECT are similar between twice and thrice a week session, but twice a week sessions are associated with fewer cognitive side effects. Depression symptoms will be assessed with the Inventory for Depressive Symptoms. Response and remission will follow standard definition of decrease ≥50% (response) and IDS < 10 (remission). Patients will receive a maximum of 16 treatments. This maximum treatment number was chosen as the number of ECT treatments for an index course in depression is 12, but available data on MST indicates that MST may require more treatment sessions to achieve remission.

Aim 1. To evaluate the feasibility of using MST to treat dPD in preparation for a future definite superiority trial comparing active MST vs. sham MST for depression in Parkinson's disease.

Hypothesis 1a: Enrollment will be ≥70% of the planned target (i.e. 14 out of 20 participants).

Hypothesis 1b: Retention rate of randomized participants will be ≥70%.

Aim 2. To characterize the side effect profile of MST in dPD, with particular emphasis on cardiovascular and cognitive side effects.

Hypothesis 2a: Drop out rates due to side effects during treatment will be ≤10%

Aim 3: To obtain mean, SD, and 95% confidence intervals of potential outcome variables for the future RCT to estimate the sample size of the future RCT.

Aim 4: To explore the use of EEG as a biomarker of treatment response and correlate of response to MST

ELIGIBILITY:
Inclusion Criteria:

1. Are outpatient or inpatient persons capable of providing informed consent;
2. ≥50 years old;
3. Confirmed diagnosis of Parkinson's disease based on UK Brain Bank criteria;
4. Hoehn and Yahr stage between 1-4;
5. MINI International Neuropsychiatric Interview diagnosis, Version 6 (MINI-6.0.) diagnosis of a current major depressive episode;
6. IDS score of ≥22 (moderate/severe depression);
7. Are on stable doses of psychotropic medication;
8. Are considered to be appropriate to receive convulsive therapy as assessed by an attending psychiatrist and a consultant anaesthesiologist;
9. Patient may or may not be on antidepressant medication, but If on antidepressant medication, they should be agreeable to keep their current antidepressant treatment constant during the intervention;
10. are able to adhere to the intervention schedule;
11. meet the MST safety criteria;

Exclusion Criteria:

1. Current diagnosis of major neurocognitive disorder other than PD (eg. Multiple System Atrophy, Lewy Body Dementia) or dementia (Montreal Cognitive Assessment (MoCA) <21)
2. Current active psychosis;
3. Have any of the cardiovascular risk factors listed on the Revised Cardiac Risk Index Score
4. Unstable medical conditions that, in the opinion of the Principal Investigator, carries significant risk of exacerbation by either of the study interventions;
5. Psychotropic medication initiation <4 weeks prior to enrolment (two classes, antiparkinsonsian and antidepressant compounds);
6. Have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
7. Require a benzodiazepine dose > 2mg/day of lorazepam or equivalent dose or are on any anticonvulsant due to the potential of these medications to limit the efficacy of MST;
8. Are unable to communicate in English fluently enough to complete the neuropsychological tests;
9. Have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).
10. Have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using MST to treat dPDT for depression in Parkinson's disease: recruitment | 18 months
  Enrollment will be ≥70% of the planned target.
Feasibility of using MST to treat dPDT for depression in Parkinson's disease: retention | 18 months
  Retention rate of randomized participants will be ≥70%
Feasibility of using MST to treat dPDT for depression in Parkinson's disease: side effects | 18 months
  Drop out rates due to side effects will be ≤10%

SECONDARY OUTCOMES:
Efficacy information to plan future definite trial | 18 months
  To obtain mean, SD, and 95% confidence intervals of potential outcome variables for the future RCT to estimate the sample size of the future RCT.
  Inventory of Depressive Symptoms (IDS-30), Quick Inventory of Depressive Symptomatology (QIDS), and MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No